CLINICAL TRIAL: NCT03584880
Title: Effect of Diode Laser Disinfection on Postoperative Pain in Retreatment Cases
Brief Title: Postoperative Pain After Root Canal Disinfection Via Diode Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ozgur Genc Sen, Assistant professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.YYU.0.01.00.00/124
Record Dates: First submitted 2018-05-29; First posted 2018-07-12 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Root Canal Infection; Pain
Keywords: postoperative pain; Diode laser; retreatment
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Diode Laser disinfection (Experimental): Diode laser disinfection Laser type: 940 nm diode laser Power: 1 Watt Tip: 200 micrometer fibre tip
  Interventions: Device: Diode laser disinfection
- Pseudo Diode Laser Disinfection (Placebo Comparator): Inactivated Diode laser application in root canal
  Interventions: Device: Pseudo diode laser disinfection

INTERVENTIONS:
Device: Diode laser disinfection — Root canal disinfection using a 940 nm dental laser after the removal of root canal filling of failed endodontic cases.
  Arms: Diode Laser disinfection
Device: Pseudo diode laser disinfection — Without activating laser energy, same procedure as experimental group was performed (Sham laser application)
  Arms: Pseudo Diode Laser Disinfection

SUMMARY:
The prevention and control of post-treatment pain is of great importance for the comfort of the patient as well as for the clinician's prestige. In this study, the effect of 940 nm diode laser disinfection on the postoperative pain of retreatment cases was evaluated.

DETAILED DESCRIPTION:
From the fact that microorganisms are the most common factors causing pain, this study aimed to evaluate effect of 940 nm diode laser disinfection performed in addition to conventional irrigation on postoperative pain of retreatment cases. Eighty-four patients with chronic apical periodontitis were treated. Root canal fillings were removed using rotary files. Root canals were irrigated using sodium hypochlorite between instrument changes. Final irrigation was performed using sodium hypochlorite and ethylenediaminetetraacetic acid (EDTA). The cases were randomly allocated into 2 groups: Group 1: Diode laser disinfection group, Group 2: control group. Root canal fillings were applied and crowns were restored. All treatments were completed in a single appointment. Patients were given a pain scale and they were requested to mark the code that reflects their pain intensity during 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Only asymptomatic single rooted teeth that had an initial root canal filling diagnosed with chronic periodontitis (minimum size 2x2 mm)

Exclusion Criteria:

* teeth with root canal fillings newer than 4 years, overfilled teeth, teeth with intraradicular posts, existence of a sinus tract, consumption of antibiotics within 1 month, consumption of analgesics in last 5 days, systemic disease, pregnancy, history of trauma, traumatic occlusion

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Post-endodontic pain after diode laser disinfection in retreatment cases | 24 hours postoperatively
  Pain intensity was evaluated at 24 hours after retreatment procedures. An 11-item numerical rating scale (NRS) was used to assess the pain. This NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 -10 integers) that best reflects the intensity of their pain. Number 0 represents 'no pain' whereas number 10 represents 'pain as bad as someone can imagine'.All patients were requested to mark a number corresponding to their average pain.

SECONDARY OUTCOMES:
Post-endodontic pain after diode laser disinfection in retreatment cases | 24 to 48 hours postoperatively
  Pain intensity was evaluated at 48 hours after retreatment procedures. An 11-item numerical rating scale (NRS) was used to assess the pain. This NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 -10 integers) that best reflects the intensity of their pain. Number 0 represents 'no pain' whereas number 10 represents 'pain as bad as someone can imagine' . All patients were requested to mark a number corresponding to their average pain.
Post-endodontic pain after diode laser disinfection in retreatment cases | 48 to 72 hours postoperatively
  Pain intensity was evaluated at 72 hours after retreatment procedures. An 11-item numerical rating scale (NRS) was used to assess the pain. This NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 -10 integers) that best reflects the intensity of their pain. Number 0 represents 'no pain' whereas number 10 represents 'pain as bad as someone can imagine'. All patients were requested to mark a number corresponding to their average pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur Genc Sen, Principal Investigator — Yuzuncu Yil University, Faculty of Dentistry; Melih Kaya, PhD, Study Director — Yuzuncu Yıl University, Faculty of Dentistry
Locations (1):
- Ozgur Genc Sen, Van, Türkiye (tur), Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Genc Sen O, Kaya M. Effect of Root Canal Disinfection with a Diode Laser on Postoperative Pain After Endodontic Retreatment. Photobiomodul Photomed Laser Surg. 2019 Feb;37(2):85-90. doi: 10.1089/photob.2018.4539. Epub 2019 Jan 14. PMID 31050927